CLINICAL TRIAL: NCT02368938
Title: Prognosis Factors of Mortality and Cardiovascular Diseases in the Elderly Chinese: the Northern Shanghai Study
Brief Title: Prognosis in the Elderly Chinese: the Northern Shanghai Study
Acronym: NSS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Professor in medicine, clinical chief, Shanghai 10th People's Hospital
Other Study IDs: NSS
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Risk Factor
Keywords: Cardiovascular risk factors; Prospective study; Mortality; Cardiovascular events; Asymptomatic target organ damage; elderly Chinese

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pasting venous blood sample and urine sample were collected for each participant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Several communities in the north of Shanghai

SUMMARY:
The Northern Shanghai Study is a prospective community-based study, which is aimed to investigate the prognostic factors, including conventional cardiovascular risk factors and asymptomatic target organ damage, for mortality and cardiovascular diseases, in 5,000 elderly Chinese.

ELIGIBILITY:
Inclusion Criteria:

1. age≥65 years old(depending on identity card);
2. informed consent should be signed voluntarily;
3. the individuals are long-term residents in northern Shanghai.

Exclusion Criteria:

1. is diagnosed serious heart disease (NYHA>IV) or end stage renal disease (CKD > 4);
2. suffered with cancer and life expectancy was less than 5 years;
3. has stroke within 3 months;
4. is not willing to participate in the clinical study;
5. suffered with other disease to quite the trial;
6. violated the protocol;
7. lost contact with laboratory staff.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 5000 subjects aged over 65 years old, living in communities located in the northern Shanghai, will be invited to participate in the present study, if they are willing to give their written informed consents.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
all-cause and cardiovascular mortality, cardiovascular events | one year
Cardiovascular diseases | one year

REFERENCES:
- [Derived] Han J, Tang J, Zhao Y, Xiong J, Zhao S, Yue W, Xu Y, Yu S, Zhang Y; Northern Shanghai Study. Subendocardial Viability Ratio Is Associated With Target Organ Damage and Hints at a Potential Independent Predictor of Cardiovascular Mortality in Older Adults: A Prospective Cohort Study. J Am Heart Assoc. 2026 Jan 6;15(1):e043643. doi: 10.1161/JAHA.125.043643. Epub 2025 Dec 30. PMID 41467407
- [Derived] Xu C, Zhao S, Tang J, Han J, Zhang H, Liu W, Zhao Y, Xu Y, Zhang Y. Associations between different anthropometric measures and major adverse cardiovascular events among the elderly in China. Obes Res Clin Pract. 2025 Nov-Dec;19(6):497-502. doi: 10.1016/j.orcp.2025.10.010. Epub 2025 Nov 9. PMID 41207843
- [Derived] Shi J, Ye X, Yu S, Zhao Y, Xiong J, Ji H, Zhang Y. Vascular Aging, Cardiovascular-Kidney-Metabolic Syndrome, and Cardiovascular Risk: The Northern Shanghai Study. JACC Adv. 2025 Oct 16;4(12):102242. doi: 10.1016/j.jacadv.2025.102242. Online ahead of print. PMID 41165644
- [Derived] Ren Z, Yang H, Zhu W, Han J, Yu S, Zhao S, Meng W, Xu Y, Zhao Y, Zhang Y. Age and blood pressure stratified healthy vascular aging, organ damage and prognosis in the community-dwelling elderly: insights from the North Shanghai Study. Clin Hypertens. 2024 Nov 1;30(1):31. doi: 10.1186/s40885-024-00288-3. PMID 39482774
- [Derived] Zhao S, Tang J, Yu S, Maimaitiaili R, Teliewubai J, Xu C, Li J, Chi C, Xu Y, Zhang Y. Monocyte to high-density lipoprotein ratio presents a linear association with atherosclerosis and nonlinear association with arteriosclerosis in elderly Chinese population: The Northern Shanghai Study. Nutr Metab Cardiovasc Dis. 2023 Mar;33(3):577-583. doi: 10.1016/j.numecd.2022.12.002. Epub 2022 Dec 10. PMID 36646605
- [Derived] Lyu Y, Yu S, Chi C, Teliewubai J, Li J, Blacher J, Pu J, Zhang Y, Xu Y. Associations of Walking Activity With Hypertensive Mediated Organ Damage in Community-Dwelling Elderly Chinese: The Northern Shanghai Study. Front Cardiovasc Med. 2021 Oct 21;8:734766. doi: 10.3389/fcvm.2021.734766. eCollection 2021. PMID 34746252
- [Derived] Ren Z, Zhang J, Yu S, Zhao S, Tang J, Zheng Y, Meng W, Xu C, Zhang Y, Xu Y. Hypertension-Mediated Organ Damage Correlates With Serum Homocysteine Level in Community-Dwelling Elderly Chinese: The North Shanghai Study. Front Cardiovasc Med. 2021 May 10;8:662741. doi: 10.3389/fcvm.2021.662741. eCollection 2021. PMID 34041284
- [Derived] Xu C, Zhao S, Yu S, Chi C, Fan X, Ji H, Maimaitiaili R, Teliewubai J, Li X, Zhang Y, Xu Y. Association between organ damage and visceral adiposity index in community-dwelling elderly Chinese population: the Northern Shanghai Study. Aging Clin Exp Res. 2021 Aug;33(8):2291-2297. doi: 10.1007/s40520-020-01752-4. Epub 2020 Nov 21. PMID 33219935
- [Derived] Teliewubai J, Fan X, Ji H, Maimaitiaili R, Tang J, Zhao S, Yu S, Chi C, Xu Y, Zhang Y. Does healthy obesity exist in the elderly? Findings from the Northern Shanghai Study. Nutr Metab Cardiovasc Dis. 2020 May 7;30(5):749-757. doi: 10.1016/j.numecd.2020.01.010. Epub 2020 Jan 25. PMID 32249139
- [Derived] Fan X, Teliewubai J, Xiong J, Chi C, Lu Y, Zhu M, Zhang Y, Xu Y. Renal functional impairment in the elderly, the importance of fasting plasma glucose: the Northern Shanghai Study. Aging Clin Exp Res. 2021 Feb;33(2):353-360. doi: 10.1007/s40520-020-01527-x. Epub 2020 Mar 21. PMID 32200498
- [Derived] Chi C, Teliewubai J, Lu YY, Fan XM, Yu SK, Xiong J, Zhou YW, Ji HW, Zhang Y, Xu YW. Comparison of various lipid parameters in association of target organ damage: a cohort study. Lipids Health Dis. 2018 Aug 25;17(1):199. doi: 10.1186/s12944-018-0800-y. PMID 30144803
- [Derived] Teliewubai J, Bai B, Zhou Y, Lu Y, Yu S, Chi C, Li J, Blacher J, Xu Y, Zhang Y. Association of asymptomatic target organ damage with secreted frizzled related protein 5 in the elderly: the Northern Shanghai Study. Clin Interv Aging. 2018 Mar 6;13:389-395. doi: 10.2147/CIA.S155514. eCollection 2018. PMID 29551893
- [Derived] Xiong J, Yu X, Yu S, Bai B, Xu H, Ji H, Teliewubai J, Wang K, Chi C, Lu Y, Zhou Y, Fan X, Li J, Zhang Y, Xu Y. Comparison of central and peripheral hemodynamics in association with left ventricular diastolic dysfunction in the community-based elderly Chinese. J Am Soc Hypertens. 2017 Jun;11(6):366-375. doi: 10.1016/j.jash.2017.04.009. Epub 2017 Apr 27. PMID 28528875
- [Derived] Ji H, Xiong J, Yu S, Chi C, Fan X, Bai B, Zhou Y, Teliewubai J, Lu Y, Xu H, Zhang Y, Xu Y. Northern Shanghai Study: cardiovascular risk and its associated factors in the Chinese elderly-a study protocol of a prospective study design. BMJ Open. 2017 Mar 29;7(3):e013880. doi: 10.1136/bmjopen-2016-013880. PMID 28360242
- [Derived] Lu Y, Zhu M, Bai B, Chi C, Yu S, Teliewubai J, Xu H, Wang K, Xiong J, Zhou Y, Ji H, Fan X, Yu X, Li J, Blacher J, Zhang Y, Xu Y. Comparison of Carotid-Femoral and Brachial-Ankle Pulse-Wave Velocity in Association With Target Organ Damage in the Community-Dwelling Elderly Chinese: The Northern Shanghai Study. J Am Heart Assoc. 2017 Feb 20;6(2):e004168. doi: 10.1161/JAHA.116.004168. PMID 28219916